CLINICAL TRIAL: NCT05491278
Title: Efficacy and Safety of Fospropofol Disodium Versus Propofol for Sedation in Mechanically Ventilated ICU Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xiaobo Yang, MD (Other)
Responsible Party: Sponsor-Investigator, Xiaobo Yang, MD, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WUHICU202206
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-09

CONDITIONS: Critical Illness
Keywords: Fospropofol; Propofol; Sedation; Intensive care unit
MeSH Terms: conditions — Critical Illness | interventions — fospropofol; Injections; Remifentanil; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fospropofol disodium for injection (Experimental): Fospropofol disodium continuous infusion to reach a RASS score of -3 to 0. Remifentanil continuous infusion of 4 to 9 ug/kg/h for analgesia.The dosage adjustment plan was determined by the attending physician. Whether to use other sedative drugs is up to the attending physician.
  Interventions: Drug: Fospropofol disodium for injection
- propofol (Active Comparator): Propofol continuous infusion to reach a RASS score of -3 to 0. Remifentanil continuous infusion of 4 to 9 ug/kg/h for analgesia. The dosage adjustment plan was determined by the attending physician. Whether to use other sedative drugs is up to the attending physician.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Fospropofol disodium for injection — Fospropofol disodium for injection continuous infusion to reach a RASS score of -3 to 0. Remifentanil continuous infusion of 4 to 9 ug/kg/h for. The dosage adjustment plan was determined by the attending physician. Whether to use other sedative drugs is up to the attending physician.
  Other Names: Remifentanil
  Arms: Fospropofol disodium for injection
Drug: Propofol — Propofol for injection continuous infusion to reach a RASS score of -3 to 0. Remifentanil continuous infusion of 4 to 9 ug/kg/h for. The dosage adjustment plan was determined by the attending physician. Whether to use other sedative drugs is up to the attending physician.
  Other Names: Remifentanil
  Arms: propofol

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of fospropofol disodium for injection compared to propofol for sedation in mechanically ventilated ICU patients.

DETAILED DESCRIPTION:
This is a randomized, open-label, small sample study using fospropofol disodium and propofol for sedation in mechanically ventilated ICU patients. Subjects are randomized to different treatment groups (including 1 for fospropofol disodium and 1 for propofol). Remifentanil is co-administered with fospropofol or propofol. Efficacy and safety profiles of fospropofol disodium are to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >= 18 and <= 75 years; Endotracheal intubated; Patients currently on mechanical ventilation <= 96 hours and expected to be mechanically ventilated >= 24 hours; Demand for light/moderate sedation (a RASS score of -3 to 0).

Exclusion Criteria:

* Informed Consent is unsigned； Participated in any other interventional research within 3 months; Tracheostomy; BMI <= 18 and >= 35 kilograms per square meter Pregnant; Lactant; Known or suspected allergy to various components of the study drug or to opioids and their salvage drugs, or other diseases (such as pancreatitis associated with hyperlipidemia) for which lipid emulsion should not be used; Patients who cannot be evaluated for RASS for various reasons (such as mental illness, acquired or congenital mental retardation, deafness, severe neuromuscular disease, Parkinson's disease, Huntington's disease, Alzheimer's disease, cerebrovascular disease, coma, or severe cognitive impairment due to structural diseases such as stroke, intracranial hemorrhage, head injury, malignancy, hypoxic brain injury, or cerebral edema); Patients with an expected survival period of less than 48 hours; Severe hepatic insufficiency (CTP score is 10-15 points); Chronic kidney disease (CKD grade 3 above); Unstable angina pectoris or acute myocardial infarction; Left ventricular ejection fraction <= 30%; Heart rate < 50bpm(intravenous pumping of isoproterenol <4ug/min, heart rate ≥50bpm may not be excluded); Type 2 second-degree or third-degree atrioventricular block (except those implanted a pacemaker); Two vasoconstrictors are used to maintain SBP above 90mmHg after sufficient fluid resuscitation; Myasthenia gravis; Patients with a history of drug abuse, drug abuse, alcohol abuse and long-term use of psychotropic drugs within 2 years before the screening period. Binge drinking is defined as regular drinking more than 14 times per week (1 time = 150ml of wine or 360ml of beer or 45ml of spirits);

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent reaching sedation goals | Within 7 days of the study began
  Proportion of RASS assessment time points for subjects meeting target sedation levels among all RASS assessment time points during study drug administration without rescue sedation.

SECONDARY OUTCOMES:
Invasive ventilator free time within 7 days | Within 7 days of the study began
  The time without invasive ventilation within 7 days of the study began
Rate of successful extubation within 7 days | Within 7 days of the study began
  The proportion of participants who experienced successful extubation within 7 days of the study began
Incidence of unexpected extubation | Within 7 days of the study began
  Incidence of all extubation not planned by the attending physician
Proportion of delirium in the ICU | During ICU stay
  Delirium as a percentage of all evaluable mental patients in the ICU
Non-ICU survival time within 28 days | Within 28 days of the study began
  The time of survival outside of ICU within 7 days of the study began
Case fatality rate within 28 days | Within 28 days of the study began
  After follow-up, the fatality rates of all enrolled patients (including those still in ICU, transferred out and discharge) within 28 days of the study began
Percentage of time spent that trial drug was discontinued due to adverse events | Within 7 days of the study began
  Percentage of time the trial drug was discontinued due to any adverse event suspected to be related to the trial drug

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care Medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China

IPD SHARING:
Plan to Share IPD: Undecided